CLINICAL TRIAL: NCT01037387
Title: Effect of the Noninvasive Mechanical Ventilation on the Daily Physical Activity and the Inflammatory Biomarkers in Stable Patients With COPD
Brief Title: Effect of Noninvasive Ventilation on Physical Activity and Inflammation in COPD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP PI-825
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia | interventions — Bronchodilator Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Conventional treatment for COPD
  Interventions: Drug: Control
- NIMV group (Experimental): NIMV: Conventional treatment plus noninvasive mechanical ventilation
  Interventions: Device: NIMV group

INTERVENTIONS:
Drug: Control — Current treatment according to the ATS/ERS guidelines
  Other Names: Bronchodilator agents and inhaled corticosteroids
  Arms: Control
Device: NIMV group — Current treatment according to the ATS/ERS guidelines and nocturnal BiPAP (IPAP 10-20 cmH2O,EPAP 4-6 cmH2O).
  Other Names: Bronchodilator agents and inhaled corticosteroids.
  Arms: NIMV group

SUMMARY:
Parallel, randomized and controlled clinical trial to evaluate the effect of 12 months of noninvasive mechanical ventilation versus conventional treatment in hypercapnic patients with stable COPD.

Main objective: To evaluate the effect of 12 months of noninvasive ventilation on c-reactive protein concentration and daily physical activity in hypercapnic patients with stable COPD.

Secondary objectives: To compare the plasmatic concentration of other inflammatory biomarkers between COPD patients with conventional treatment and wich noninvasive ventilation. To determine the response of breathlessness, health-related quality of life and lung function to noninvasive ventilation. To identify the COPD patients with a higher gasometric and clinic response to noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-75 yrs.
* COPD diagnosis (postbronchodilator FEV1/FVC < 0.7) for at least 6 months.
* FEV1 < 45% predicted
* Baseline pH 7.35-7.45
* Baseline PaCO2>45 mmHg breathing current air
* Smoking history (>15 pack-year)
* Clinically stable for at least the last three months
* Pharmacological treatment optimized in the last two years.

Exclusion Criteria:

* Previous diagnosis of asthma, other airway obstructive disease, sleep apnea syndrome, interstitial lung disease, chest wall disease or neuromuscular disease.
* Apnea-hypopnea index > 10/h
* Morbid obesity (BMI > 45 Kg/m2)
* Previous diagnosis of ischaemic heart disease, cardiac failure, cirrhosis, chronic renal failure, rheumatoid arthritis or other inflammatory disease.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
daily physical activity and plasmatic concentration of C-reactive protein | 12 months

SECONDARY OUTCOMES:
Seric concentrations of homocysteine, proBNP, fibrinogen, cholesterol, tg, tnf-alpha, IL-1, IL-6 and 8-isoprostane | 12 months
PaO2, PaCO2, pH, IC, VCIN, FVC, FEV1, FEV1/FVC, TLC, FRC/TLC, RV/TLC,PImax, PEmax, TTmus, 6MWD | 12 months
BDI/TDI, SF-36, SGRQ, LCADL | 12 months
Adverse effects | 12 months
Cardiovascular effects, exacerbations, hospitalizations and mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonia Gómez-Mendieta, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain